CLINICAL TRIAL: NCT01108354
Title: The Serotonin Transporter in Attention Deficit Hyperactivity Disorder Investigated With Positron Emission Tomography
Brief Title: The Serotonin Transporter in Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof. PD Dr., Medical University of Vienna
Other Study IDs: AP13675ONB
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD patients: 10 male adult ADHD patients and 10 female adult ADHD patients
- healthy controls: 20 age- and sex-matched healthy volunteers

SUMMARY:
The aim of the present proposal is to prove that adult attention deficit hyperactivity disorder (ADHD) patients show lower serotonin transporter (5-HTT) binding using positron emission tomography (PET) and the selective radioligand [11C]DASB. Specifically, the 5-HTT binding will be quantified in 20 adult medication-free ADHD patients (50% females) and in 20 age- and sexmatched healthy controls. Investigating untreated adult ADHD patients without any psychiatric comorbidities will provide the opportunity to estimate the change of serotonin transporter binding in adult ADHD patients compared to a group of healthy controls. Several lines of evidence support the hypothesis that serotonergic neurotransmission may, in addition to dopamine, play an important role in the aetiology of ADHD. So far, no PET study investigating serotonergic neurotransmission in adult ADHD patients has been conducted, although alterations in the serotonin system may be substantially involved in the susceptibility and subtype characterization of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female outpatients who are at least 18 years of age and no more than 65 years of age when informed consent is obtained.
* Patients must meet DSM-IV-TR criteria for current ADHD as well as for historical diagnosis of ADHD during childhood as assessed by the Conner´s Adult ADHD Diagnostic Interview for DSM-IV (CAADID, Conners 1999).
* Patients must have a score of >2 on at least 6 items of either the inattentive or hyperactive score subscales at screening on the rated CAARS-Inv:SV (Conners 1999). In addition, their CAARS-Inv:SV 18-item total ADHD symptom score (the sum of the inattention and hyperactivity/impulsivity subscales) must be >20.
* Patients must have a CGI-ADHD-S score of >4 (moderate symptoms) at screening.
* Patients must be physically healthy.
* Patients must be able to understand and willing to sign the written informed consent document.

Exclusion Criteria:

* Patients suffering from severe somatic diseases will be excluded from the study.
* Any treatment with stimulants, selective norepinephrine reuptake inhibitors or any other psychotropic treatments, such as SSRIs, etc. within six months prior to screening.
* Patients suffering from any current comorbid psychiatric disorder (Axis I or Axis II diagnosis according to DSM-IV-TR) will be excluded.
* Patients who are currently using alcohol, drugs of abuse, or any medication in a manner which is indicative of chronic abuse or who meet DSM-IV-TR criteria for alcohol or other substance dependence.
* Any implant or stainless steel graft.
* Positive urine pregnancy test.
* Participation in studies with PET or SPECT within the last 10 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 participants including ten male adult ADHD patients, ten female adult ADHD patients and 20 age- and sex-matched healthy volunteers, free of any psychotropic treatments at baseline
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
5-HTT-binding potential | 16 months
  5-HTT-binding potential in adult medication-free ADHD patients compared to a group of healthy controls

SECONDARY OUTCOMES:
SNPs | 16 months
  Single nucleotide polymorphisms (SNPs)of three genes, the serotonin transporter gene (SLC6A4), the 5-HT1A receptor gene[(-1018)G>C], and the 5-HT2A receptor gene [102T/C]

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mitterhauser, PhD A/Prof, Principal Investigator — Medical University of Vienna; Alexandra Kutzelnigg, MD, Principal Investigator — Medical University of Vienna; Rupert Lanzenberger, MD. A/Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.meduniwien.ac.at/neuroimaging/